CLINICAL TRIAL: NCT00175370
Title: Treatment of Catheter Related Bloodstream Infection Caused by Coagulase Negative Staphylococcus; Removal of Catheter Followed by 2 Days Compared With 7 Days Intravenous Vancomycin
Brief Title: Vancomycin Study: Treatment of Catheter Related Bloodstream Infection Caused by Coagulase Negative Staphylococcus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Jane de Lemos, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C00-0106
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Staphylococcal Infections
Keywords: Vancomycin; Coagulase Negative Staphylococcus; Central Venous Catheter; Bloodstream infection; CNS bloodstream infection
MeSH Terms: conditions — Staphylococcal Infections; Sepsis | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vancomycin — Randomized double-blind equivalence trial to test the hypothesis that 2 days is equivalent to 7 days of vancomycin treatment for intravascular device associated bacteremia due to coagulase negative staphylococcus. The definitions for the surveillance of intravascular device associated bacteremia from the Laboratory Centre for Disease Control-Health Canada will be used. Surveillance blood cultures on days 4 and 9 following removal of intravascular device. Relatedness of strains will be determined by pulsed-field gel electrophoresis (PFGE).

SUMMARY:
Patients admitted into the Intensive Care Unit (ICU) have an intravenous (IV) catheter (small plastic tube) placed in their vein. Very occasionally (4 times out of 100) the insertion of an intravenous catheter may cause an infection in the blood. It has been shown that the removal of the catheter and the insertion of a new one at a new site helps to get rid of this infection. Sometimes, antibiotics are also given.

Vancomycin is the antibiotic given intravenously (into the vein) to treat these catheter-related infections. At Vancouver General Hospital, some physicians may not give any vancomycin at all whereas others may treat with intravenous (IV) vancomycin for one to fourteen days.

Since there are a lack of data to support the length of IV vancomycin therapy, the investigators would like to find out if two days of IV vancomycin are as good as seven days.

Therefore, the purpose of this study is to determine if two days of IV vancomycin are as good as seven days for the treatment of catheter-related infections in the blood.

DETAILED DESCRIPTION:
INTRODUCTION: Intravascular device associated bacteremia due to coagulase negative staphylococcus has become the most common nosocomial bacteremia. Despite its prevalence, no prospective study has investigated how these infections should be treated. Removal of the intravascular device is associated with a reduction in recurrence rate from 20% to 3% but the required duration of vancomycin therapy is not known. We propose to test the hypothesis that, following removal of the intravascular device, treatment with 2 days of vancomycin is equivalent to 7 days of vancomycin.

INTERVENTION: Randomized double-blind equivalence trial to test the hypothesis that 2 days is equivalent to 7 days of vancomycin treatment for intravascular device associated bacteremia due to coagulase negative staphylococcus. The definitions for the surveillance of intravascular device associated bacteremia from the Laboratory Centre for Disease Control-Health Canada will be used.

MEASUREMENTS: Surveillance blood cultures on days 4 and 9 following removal of intravascular device. Relatedness of strains will be determined by pulsed-field gel electrophoresis (PFGE).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU who require treatment for suspected or documented intravascular device associated (IVDA) bacteremia due to coagulase-negative staphylococci (CNS). Suspected IVDA bacteremia due to CNS is defined as finding of gram positive cocci in blood in a patient with either an intravascular device (IVD) in situ or within 24 hours of catheter removal, with clinical signs of sepsis:

  * two signs of systemic inflammatory response syndrome (SIRS): heart rate (HR) > 90, Temp > 38 or < 36, white blood cell (WBC) > 12 or < 4, respiratory rate (RR) > 20 or pCO2 < 32; and
  * with no obvious source of bacteremia other than the IVD.

Exclusion Criteria:

* Underlying valvular heart disease
* Prosthetic valve or graft
* A history of infectious endocarditis
* Bone marrow transplant recipient
* Neutropenia (< 0.5 X 10^9/L)
* Solid organ transplant recipient
* Known hypersensitivity to vancomycin
* Calculated creatinine clearance < 25 ml/min

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2000-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement will be the proportion of patients with early bacteriological failure | Nine days
Early bacteriologic failure | Nine days
Recovery in blood culture of an isolate with same antibiogram, biotype and PFGE type as the initial bacteria, from any blood culture, up to 9 days following IVD removal | Nine days

SECONDARY OUTCOMES:
The secondary endpoint will be the proportion of patients with clinical failure, late bacteriologic failure and recurrent bacteremia. | Nine days

CONTACTS AND LOCATIONS:
Overall Officials: Jane de Lemos, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital Intensive Care Unit, Vancouver, British Columbia, Canada